CLINICAL TRIAL: NCT00428662
Title: Clinical and Angiographic Evaluation of Paclitaxel Eluting, Non-Polymeric, Nanoporous Carbon-Carbon Coated, Cobalt-Chromium Stent
Brief Title: Evaluation of a New Nanotechnology Based Drug-Eluting Stent for Opening of Narrowed Arteries of the Heart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0101
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2007-01-30 (Estimated); Status verified 2007-01

CONDITIONS: Coronary Stenosis
Keywords: coronary stenting; drug eluting stents; paclitaxel; nanoporous
MeSH Terms: conditions — Coronary Stenosis

INTERVENTIONS:
Device: drug eluting nonpolymeric nanoporous stent

SUMMARY:
Coronary artery disease (CAD) is the largest cause of death and disability in the world. Besides medicines, the principle treatment of this condition requires opening of the narrowed arteries, responsible for angina and other symptoms of the disease, by angioplasty or surgery. Introduction of metal scaffolds called 'stents' in the past few decades revolutionised the angioplasty technique, and has made it the most popular treatment today for CAD. However these stents are prone to becomin narrow and obstructed after implanataion, causing symptoms and non-fatal heart attacks in some patients. Introduction of stents that slowly release drugs locally to minimize this process, called 'drug-eluting stents'(DES)he past few years has been one of the biggest breakthroughs in the field of cardiology. However ven the current available DES are still prone to narrowing in high-risk patients, like those with diabetes, and also have a higher chance for sudden blockage by a blood clot even many years later after insertion. Thus it is important to develop technology for more efficacious and safer DES.This includes safer drugs, better stent design and delivery, and more inert platforms for drug release We hypothesise that a new stent made with nanoporous particle with better polymer for drug release will prove to be safer and more efficacious alternative to currently available DES.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female 2: 18 years of age (note: females of child bearing potential must have a negative pregnancy test within 7 days of treatment and must use effective pregnancy avoidance until the 6 month angiogram is completed)
2. Have chest pain consistent with angina pectoris or a history of documented myocardial infarction or documented silent ischemia
3. Treatment of a native vessel de novo coronary lesion (only 1 single study lesion/patient)
4. Target vesseI2.5mm-4.0mm in diameter (visual estimate)
5. Target lesion length::: 12mm (visual estimate)
6. Target lesion stenosis> 50% and < 100% (visual estimate)
7. At least TIMI grade II coronary flow
8. Acceptable candidate for CABG surgery
9. Patient is willing to come back for a follow-up evaluations including repeat cardiac catheterization 5-7 months after treatment
10. Patient must provide written informed consent prior to the index procedure using a form that is approved by the local Ethics Committee

Exclusion Criteria:

1. Patient has experienced an acute myocardial infarction (Q wave or non-Q wave) within 72 hours prior to the index procedure with CK enzymes 2: 2x the local laboratory upper limit of normal, with the presence of CK- MB levels elevated above the local laboratory upper limit of normal;
2. Unprotected left main coronary disease with> 50% stenosis;
3. Significant (> 50%) stenosis proximal or distal to the target lesion that might require revascularization or impede runoff;
4. Ostial location of the target lesion;
5. Angiographic evidence of thrombus within the target lesion;
6. Severely calcified'lesion which cannot be successfully predilated;
7. Documented L VEF < 25%, or clinically significant congestive cardiac failure;
8. Totally occluded vessel;
9. Impaired renal function (creatinine> 0.27mmol/L) at the time of treatment;
10. Pretreatment with devices other than balloon angioplasty;
11. Excessive tortuosity proximal to the lesion which makes stent delivery and deployment uncertain;
12. Target lesion involves a bifurcation including a diseased side branch> 2.5mm in diameter that would require treatment;
13. Prior stenting within 5mm of the target lesion;
14. Patient is a recipient of a heart transplant;
15. Patient has a life expectancy < 12 months;
16. Known allergies to clopidogrel bisulfate (Plavix@), ticlopidine (Ticlid@), Cobalt Chromium alloy and Paclitaxol that cannot be medically managed;
17. In the investigator's opinion, any significant medical condition which may interfere with the patient's optimal participation in this study;
18. Currently participating in an investigational drug or device study that has not completed the primary endpoint;
19. Intervention of another coronary lesion has occurred within 30 days before or is planned within 30 days after the index procedure.
20. In the investigator's opinion, the lesion is not suitable for stenting

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2007-01; Study Completion 2007-10

PRIMARY OUTCOMES:
In-stent late loss as compared historically to other DES, within the stented segment post-procedure and at 6-9-month follow-up

SECONDARY OUTCOMES:
Major adverse cardiac events
Stent thrombosis rate (acute, subacute, or chornic)

CONTACTS AND LOCATIONS:
Overall Officials: Balram Bhargava, MD, DM, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Morice MC, Serruys PW, Sousa JE, Fajadet J, Ban Hayashi E, Perin M, Colombo A, Schuler G, Barragan P, Guagliumi G, Molnar F, Falotico R; RAVEL Study Group. Randomized Study with the Sirolimus-Coated Bx Velocity Balloon-Expandable Stent in the Treatment of Patients with de Novo Native Coronary Artery Lesions. A randomized comparison of a sirolimus-eluting stent with a standard stent for coronary revascularization. N Engl J Med. 2002 Jun 6;346(23):1773-80. doi: 10.1056/NEJMoa012843. PMID 12050336
- [Background] Stone GW, Ellis SG, Cox DA, Hermiller J, O'Shaughnessy C, Mann JT, Turco M, Caputo R, Bergin P, Greenberg J, Popma JJ, Russell ME; TAXUS-IV Investigators. A polymer-based, paclitaxel-eluting stent in patients with coronary artery disease. N Engl J Med. 2004 Jan 15;350(3):221-31. doi: 10.1056/NEJMoa032441. PMID 14724301
- [Background] Bhargava B, Reddy NK, Karthikeyan G, Raju R, Mishra S, Singh S, Waksman R, Virmani R, Somaraju B. A novel paclitaxel-eluting porous carbon-carbon nanoparticle coated, nonpolymeric cobalt-chromium stent: evaluation in a porcine model. Catheter Cardiovasc Interv. 2006 May;67(5):698-702. doi: 10.1002/ccd.20698. PMID 16575925
- [Background] van der Giessen WJ, Lincoff AM, Schwartz RS, van Beusekom HM, Serruys PW, Holmes DR Jr, Ellis SG, Topol EJ. Marked inflammatory sequelae to implantation of biodegradable and nonbiodegradable polymers in porcine coronary arteries. Circulation. 1996 Oct 1;94(7):1690-7. doi: 10.1161/01.cir.94.7.1690. PMID 8840862